CLINICAL TRIAL: NCT04075487
Title: Evidence-Based Multidimensional Pain Self-Management Planning: Personalized by and for Veterans Via Web-Based Application
Brief Title: MEPS-Pain: Personalized Pain Self-management Planning by and for Veterans Pilot Study
Acronym: MEPS-Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Maryland Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A3169-P; I21RX003169-01A1 (NIH)
Record Dates: First submitted 2019-06-25; First posted 2019-08-30 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Chronic Low Back Pain
Keywords: Low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Pilot study of feasibility and user experience of minimal risk App for pain self-management intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- User experiences with MEPS-Pain (Experimental): This is a pilot study to assess user experience with MEPS-Pain App, there is only one arm.
  Interventions: Other: Web-module for patient education and planning

INTERVENTIONS:
Other: Web-module for patient education and planning — Our goal is a mobile web-based application (App) that provides immediate feedback to Veterans seeking to develop their own pain self-management plan

SUMMARY:
Chronic low back pain is the #1 cause of disability and low quality of life in Veterans. Pain is a huge burden- stealing enjoyment, fulfillment, and time. Sometimes surgery, injections, or medications can help but sometimes not. Although no one solution fixes chronic low back pain, there are many treatments that can reduce pain impact and restore quality of life. These treatments involve: movement, psychology, mind-and-body therapies, sleep, and environmental factors. The challenge is how to best coordinate these treatments for chronic low back pain. The investigators have built a prototype mobile application that delivers the latest information to Veterans so they can work with healthcare providers to build their own pain self-management plans. With this new tool, the Veteran has data at hand and chooses their preferred pain self-management activities, making a coordinated plan that can be shared with their healthcare team. The investigators' goal is giving Veterans the knowledge and power to 'plan the work and work the plan' for chronic low back pain: restoring value, fulfillment, and meaning.

DETAILED DESCRIPTION:
Chronic low back pain is highly prevalent in Veterans, and is often resistant to pharmacological management so that non-pharmacological management is required. For many patients, the most effective approach is comprehensive pain management incorporating multiple therapies addressing: physical, mental, mind-body, sleep, safety, and environmental needs. The ultimate outcome is the development of a coordinated multidimensional evidence-based plan for pain self-management (C-MEPPS) tailored to each patient. This approach, while effective, is highly resource intensive and severely constrained by cost and health system factors.

The investigators' goal is a mobile web-based application (App) that provides immediate feedback to Veterans seeking to develop their own pain self-management plan. This will represent a novel, scalable, Veteran-driven solution to chronic low back pain aligned with VA strategic objectives 'online navigator tools.empowers Veterans to make decisions.' The investigators are focused on transferring knowledge about evidence-base practices into the primary care context to help Veterans and their healthcare providers manage pain effectively- before it gets worse. The investigators have already developed the App prototype utilizing User-Centered Design principles to optimize the user experience. Our first aim is to develop and pilot test a web-based App for Veterans, including older Veterans and women Veterans, designed to empower each in pain self-management planning: providing access and data-driven guidance about evidence-based multidimensional behavior change. The investigators' second aim is to gather pilot data targeting patient-centered and rehabilitative outcomes such as: increased activity, more sleep time, decreased pain interference and better quality of life; through use of the App and engagement in pain self-management planning.

This project brings together the expertise of skilled exercise physiologists, experienced pain and sleep clinical psychologists, pain specialists, clinical educators, geriatricians, women's health providers, and technology design experts to create a powerful new pipeline for knowledge transfer to patients and providers. Grounded in whole health and integrative approaches, nursing principles, pharmacy practices, physical therapy, and nutrition are also included in the App. The investigators are working as an interprofessional pain-focused team to put the best-available information about non-pharmacological treatments for pain into the hands of Veterans and their primary care providers. The investigators' vision is to improve the lives of Veterans with chronic low back pain, improving access to knowledge and resources and giving Veterans the power to plan their own path to better, more fulfilling living despite chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Veterans receiving care at the VAMHCS
* frequent or persistent low back pain (> 3 months)
* pain >4 on a 0-10 numeric rating scale
* willing to participate in trial of non-pharmacological therapies for pain
* ability to speak, read, and write as needed for study
* stable treatment

Exclusion Criteria:

* Veterans with cognitive or visual impairment limiting the ability to engage in self-directed self-management planning
* anticipated surgery or pain procedure during the expected study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth B. Hogans, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6/21/2022-7/15/2023; recruitment from medical center through clinic outreach and advertisement on research bulletin board
Period: Overall Study
Arm/Group | User Experiences With MEPS-Pain
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | User Experiences With MEPS-Pain
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 9
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.5 [55.5 to 66.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Veteran [Count of Participants; unit: Participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: Use of Tablet-based Application (App) for Creation of Pain Self-management Plan
Description: The investigators will assess user experience with the App, assessing actual use to create a pain self-management plan. Investigators will assess whether participants used the App to create a pain self-management plan on the tablet. The outcome will be the number of participants creating at least one pain self-management plan
Time Frame: 6 weeks
Population: Completed creation of a pain plan
Measure: Count of Participants; unit: Participants
Arm/Group | User Experiences With MEPS-Pain
Number analyzed (Participants) | 19
Participants | 19

2. Primary Outcome: Tablet-based Application (App) for Pain Self-management Planning: Patient Experience Via System Usability Scale
Description: The investigators will assess user experience with the App, usability with SUS, modified for App.
  Maximum score 50 (good outcome), minimum score 10 (poor outcome).
Time Frame: 6 weeks
Population: Completed system usability scale for the App
Measure: Mean (Standard Error); unit: sum score
Arm/Group | User Experiences With MEPS-Pain
Number analyzed (Participants) | 19
sum score | 39 (2.0)

3. Primary Outcome: Tablet-based Application (App) Use for Pain Self-management Planning: Total Days With Plan Accessed
Description: Total days with plan accessed in the App
  Maximum score 42 (good outcome), minimum score 0 (bad outcome).
Time Frame: 6 weeks
Population: Tablet-based application (App) use for pain self-management planning: total days with plan accessed
Measure: Mean (Full Range); unit: Days plan accessed
Arm/Group | User Experiences With MEPS-Pain
Number analyzed (Participants) | 17
Days plan accessed | 20 [0 to 38]

4. Secondary Outcome: Pain Intensity Completion
Description: DOD-VA Pain instrument
  Maximum score 10 (bad outcome), minimum score 1 (good outcome).
Time Frame: 6 weeks
Population: Pain intensity
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | User Experiences With MEPS-Pain
Number analyzed (Participants) | 19
score on a scale | 5.1 (.57)

5. Other Pre Specified Outcome: Tablet-based Application (App) Use for Pain Self-management Planning: Daily Logging of Activities
Description: Average number activities logged per day in the App during week 5
  Maximum score 12 (good outcome), minimum score 0 (bad outcome).
Time Frame: 5 weeks
Population: Average number activities logged per day in the App during week 5 on the days used
Measure: Mean (Standard Deviation); unit: number activities logged per day of use
Arm/Group | User Experiences With MEPS-Pain
Number analyzed (Participants) | 19
number activities logged per day of use | 7.2 (3.7)

6. Other Pre Specified Outcome: Pain Interference as Measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Measure
Description: Pain interference utilizing Patient-Reported Outcomes Measurement Information System (PROMIS) pain interference measure Data are reported as scores in the PROMIS standardized scale derived by summing raw scores and converting this based on published conversion tables.
  100 (bad outcome), 0 (good outcome).
Time Frame: 6 weeks
Population: Participants initiating the study and not withdrawing
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | User Experiences With MEPS-Pain
Number analyzed (Participants) | 19
score on a scale | 59.0 (7.4)

7. Other Pre Specified Outcome: Actigraph Sleep-time Percentage
Description: Actigraph sleep-time percentage - percent of time spent in sleep per adjudicated Actigraph recording
  25-30% (good outcome), <20% or >40% (bad outcome)
Time Frame: 6 weeks
Population: Week 6, final visit
Measure: Mean (Standard Deviation); unit: percent time in sleep
Arm/Group | User Experiences With MEPS-Pain
Number analyzed (Participants) | 17
percent time in sleep | 22.3 (8.7)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Adverse event collection performed at all in person visits and phone visits
Arm/Group | User Experiences With MEPS-Pain
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT04075487/Prot_001.pdf
  • Informed Consent Form (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT04075487/ICF_000.pdf